



## Evaluation the Effects of Propolis Lozenges Extract on Salivary Biomarkers and Its Effect on Oral Health Condition in (19\_24) Years Old

**NCT Number: not yet assigned** 

Date: 10 November 2024

## RESEARCH ETHICS: PATIENT CONSENT FORM

**Study Number: MUPRV0014** 

Patient Identification Number for this trial: No. 1



Title of Project: Evaluation the Effects of Propolis Lozenges Extract on

Salivary Biomarkers and Its Effect on Oral Health Condition in (19\_24) Years

Old

Principle investigator: Ahmed Salah Abdulmahdi Finjan

- I confirm that I have read and understand the information sheet dated for the above study and have had the opportunity to ask questions.
- I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected.
- I understand that sections of any of my medical notes may be looked at by responsible individuals from regulatory authorities where it is relevant to my taking part in research. I give permission for these individuals to have access to my records

| • I agree to take part in the above study. | | | |
|--------------------------------------------|------|------|-----------|
| Name of participant | Date | | Signature |
| Name of Person taking consent | | Date | Signature |